CLINICAL TRIAL: NCT01240057
Title: Randomized Trial of Fetoscopic Endoluminal Tracheal Occlusion (FETO) Versus Expectant Management During Pregnancy in Fetuses With Left Sided and Isolated Congenital Diaphragma Hernia and Severe Pulmonary Hypoplasia.
Brief Title: Tracheal Occlusion To Accelerate Lung Growth (TOTAL) Trial for Severe Pulmonary Hypoplasia
Acronym: TOTAL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Collaborators: King's College Hospital NHS Trust (UK) (Unknown); Hospital Clinic of Barcelona (Other); Hopital Antoine Beclere (Other); University Hospital, Bonn (Other); Mater Mothers' Hospital (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Ospedale Pediatrico Bambino Gesù, Rome (IT) (Unknown); Mount Sinai Hospital, Canada (Other); National Center for Child Health and Development, Tokyo (JP) (Unknown); The University of Texas Health Science Center, Houston (Other); Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Jan Deprest, MD, PhD, University Hospital, Gasthuisberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML 6277; B32220108118 (Other: UZ Gasthuisberg KU Leuven (Belgium))
Record Dates: First submitted 2010-08-04; First posted 2010-11-15 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Congenital Diseases; Diaphragmatic Hernia; Pulmonary Hypoplasia
Keywords: Isolated Congenital Diaphragmatic Hernia; Fetal Surgery; Pulmonary Hypoplasia
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Hernia, Diaphragmatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- expectant management during pregnancy (Placebo Comparator): watchful waiting during pregnancy
  Interventions: Other: watchful waiting during pregnancy
- fetal endoluminal tracheal occlusion (Experimental): fetoscopic balloon occlusion at 27 to 29+6 weeks of gestation
  Interventions: Procedure: fetal endoluminal tracheal occlusion

INTERVENTIONS:
Procedure: fetal endoluminal tracheal occlusion — percutaneous fetoscopy, positioning of endoluminal balloon at 27-30 weeks and whenever possible elective removal at 34 weeks
  Other Names: Balt Goldbal 2 balloon
  Arms: fetal endoluminal tracheal occlusion
Other: watchful waiting during pregnancy — pregnancy surveillance for fetal wellbeing, development of polyhydramnios and cervical shortening
  Arms: expectant management during pregnancy

SUMMARY:
This trial investigates whether prenatal intervention improves survival rate of fetuses with isolated congenital diaphragmatic hernia and severe pulmonary hypoplasia, as compared to expectant management during pregnancy, both followed by standardized postnatal care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more, who are able to consent
* Singleton pregnancy
* Anatomically and chromosomally normal fetus
* Left sided diaphragmatic hernia
* Gestation at randomization prior to 29 wks plus 5 d (so that occlusion is done at the latest on 29 wks plus 6 d)
* Estimated to have severe pulmonary hypoplasia, defined prenatally as: O/E LHR <25 %, irrespective of the liver position
* Acceptance of randomization and the consequences for the further management during pregnancy and thereafter.
* The patients must undertake the responsibility for either remaining close to, or at the FETO center, or being able to travel swiftly and within acceptable time interval to the FETO center until the balloon is removed.
* Intended postnatal treatment center must subscribe to suggested guidelines for "standardized postnatal treatment".
* Provide written consent to participate in this RCT

Exclusion Criteria:

* Maternal contraindication to fetoscopic surgery or severe medical condition in pregnancy that make fetal intervention risk full
* Technical limitations precluding fetoscopic surgery, such as severe maternal obesity, uterine fibroids or potentially others, not anticipated at the time of writing this protocol.
* Preterm labour, cervix shortened (<15 mm at randomization) or uterine anomaly strongly predisposing to preterm labour, placenta previa
* Patient age less than 18 years
* Psychosocial ineligibility, precluding consent
* Diaphragmatic hernia: right-sided or bilateral, major anomalies, isolated left-sided outside the O/E LHR limits for the inclusion criteria
* Patient refusing randomization or to comply with return to FETO center during the time period the airways are occluded or for elective removal of the balloon

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2011-11; Primary Completion 2020-03 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Survival at discharge from neonatal intensive care unit | at discharge from neonatal intensive care unit
  The baby can be discharged either alive (and then it qualifies as "surviving at discharge") or dead. Not discharged babies have not reached the primary endpoint.

SECONDARY OUTCOMES:
prenatal increase in lung volume after FETO | prior to balloon removal
  volume of lung after occlusion
grading of oxygen dependency | born >32 wks: between 28-56d of life; born <32wks: 36wks postmenstrual age
occurrence of pulmonary hypertension | within first weeks of life
  determined by cardiac ultrasound
number of days in Neonatal Intensive Care Unit (NICU) | within hospital stay
  As long as the baby is in the hospital, it is hospitalized either in NICU or in another, less intensive care unit.
  The number of days in NICU is an outcome variable, expressed in days.
number of days of ventilatory support | within NICU stay
presence of periventricular leucomalacia | 2 months of life
presence of neonatal sepsis, intraventricular haemorrhage, retinopathy grade III or higher | within hospital stay
number of days till full enteral feeding | within first 2 years of life
presence of gastro-esophagal reflux | at discharge
day of surgery | within hospital stay
requirement for use of patch for repair | at the time of postnatal surgery
bronchopulmonary dysplasia | with the first 8 weeks
  defined as oxygen need for at least 28 days
Need for Extracorporeal membrane oxygenation | during NICU admission
Defect size | at the time of postnatal surgery
number of days alive in case of postnatal death | during NICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Jan Deprest, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (12):
- University of Texas Health Science Center, Houston, Texas, United States
- Mater Mother's Hospital, Brisbane, Queensland, Australia
- University Hospitals Leuven, Leuven, Belgium
- Mount Sinai Hospital, Toronto, Ontario, Canada
- Hôpital Antoine Béclère, Clamart, France
- University Hospital of Bonn, Bonn, Germany
- Italy (2):
  - Ospedale Maggiore Policlinico, Milan
  - Ospedale Pediatrico Bambino Gesù, Rome
- National Center for Child Health and Development, Tokyo, Japan
- 1st Department of Obstetrics and Gynecology, Medical University of Warsaw, Warsaw, Poland
- Hospital Clinic Barcelona, Barcelona, Catalonia, Spain
- King's College Hospital, London, United Kingdom

REFERENCES:
- [Background] Jani JC, Nicolaides KH, Gratacos E, Valencia CM, Done E, Martinez JM, Gucciardo L, Cruz R, Deprest JA. Severe diaphragmatic hernia treated by fetal endoscopic tracheal occlusion. Ultrasound Obstet Gynecol. 2009 Sep;34(3):304-10. doi: 10.1002/uog.6450. PMID 19658113
- [Background] Deprest J, Breysem L, Gratacos E, Nicolaides K, Claus F, Debeer A, Smet MH, Proesmans M, Fayoux P, Storme L. Tracheal side effects following fetal endoscopic tracheal occlusion for severe congenital diaphragmatic hernia. Pediatr Radiol. 2010 May;40(5):670-3. doi: 10.1007/s00247-010-1579-9. Epub 2010 Mar 30. No abstract available. PMID 20352401
- [Background] Deprest JA, Gratacos E, Nicolaides K, Done E, Van Mieghem T, Gucciardo L, Claus F, Debeer A, Allegaert K, Reiss I, Tibboel D. Changing perspectives on the perinatal management of isolated congenital diaphragmatic hernia in Europe. Clin Perinatol. 2009 Jun;36(2):329-47, ix. doi: 10.1016/j.clp.2009.03.004. PMID 19559323
- [Background] Deprest JA, Hyett JA, Flake AW, Nicolaides K, Gratacos E. Current controversies in prenatal diagnosis 4: Should fetal surgery be done in all cases of severe diaphragmatic hernia? Prenat Diagn. 2009 Jan;29(1):15-9. doi: 10.1002/pd.2108. No abstract available. PMID 19125386
- [Background] Deprest JA, Flemmer AW, Gratacos E, Nicolaides K. Antenatal prediction of lung volume and in-utero treatment by fetal endoscopic tracheal occlusion in severe isolated congenital diaphragmatic hernia. Semin Fetal Neonatal Med. 2009 Feb;14(1):8-13. doi: 10.1016/j.siny.2008.08.010. Epub 2008 Oct 8. PMID 18845492
- [Background] Jani JC, Benachi A, Nicolaides KH, Allegaert K, Gratacos E, Mazkereth R, Matis J, Tibboel D, Van Heijst A, Storme L, Rousseau V, Greenough A, Deprest JA; Antenatal-CDH-Registry group. Prenatal prediction of neonatal morbidity in survivors with congenital diaphragmatic hernia: a multicenter study. Ultrasound Obstet Gynecol. 2009 Jan;33(1):64-9. doi: 10.1002/uog.6141. PMID 18844275
- [Background] Jani J, Nicolaides KH, Keller RL, Benachi A, Peralta CF, Favre R, Moreno O, Tibboel D, Lipitz S, Eggink A, Vaast P, Allegaert K, Harrison M, Deprest J; Antenatal-CDH-Registry Group. Observed to expected lung area to head circumference ratio in the prediction of survival in fetuses with isolated diaphragmatic hernia. Ultrasound Obstet Gynecol. 2007 Jul;30(1):67-71. doi: 10.1002/uog.4052. PMID 17587219
- [Background] Jani J, Keller RL, Benachi A, Nicolaides KH, Favre R, Gratacos E, Laudy J, Eisenberg V, Eggink A, Vaast P, Deprest J; Antenatal-CDH-Registry Group. Prenatal prediction of survival in isolated left-sided diaphragmatic hernia. Ultrasound Obstet Gynecol. 2006 Jan;27(1):18-22. doi: 10.1002/uog.2688. PMID 16374756
- [Background] Deprest J, Gratacos E, Nicolaides KH; FETO Task Group. Fetoscopic tracheal occlusion (FETO) for severe congenital diaphragmatic hernia: evolution of a technique and preliminary results. Ultrasound Obstet Gynecol. 2004 Aug;24(2):121-6. doi: 10.1002/uog.1711. PMID 15287047
- [Background] Rodrigues HC, Deprest J, v d Berg PP. When referring physicians and researchers disagree on equipoise: the TOTAL trial experience. Prenat Diagn. 2011 Jun;31(6):589-94. doi: 10.1002/pd.2756. Epub 2011 Apr 11. PMID 21484841
- [Derived] Deprest J, Flake A. How should fetal surgery for congenital diaphragmatic hernia be implemented in the post-TOTAL trial era: A discussion. Prenat Diagn. 2022 Mar;42(3):301-309. doi: 10.1002/pd.6091. Epub 2022 Jan 22. PMID 35032132
- [Derived] Van Calster B, Benachi A, Nicolaides KH, Gratacos E, Berg C, Persico N, Gardener GJ, Belfort M, Ville Y, Ryan G, Johnson A, Sago H, Kosinski P, Bagolan P, Van Mieghem T, DeKoninck PLJ, Russo FM, Hooper SB, Deprest JA. The randomized Tracheal Occlusion To Accelerate Lung growth (TOTAL)-trials on fetal surgery for congenital diaphragmatic hernia: reanalysis using pooled data. Am J Obstet Gynecol. 2022 Apr;226(4):560.e1-560.e24. doi: 10.1016/j.ajog.2021.11.1351. Epub 2021 Nov 19. PMID 34808130
- [Derived] Deprest JA, Nicolaides KH, Benachi A, Gratacos E, Ryan G, Persico N, Sago H, Johnson A, Wielgos M, Berg C, Van Calster B, Russo FM; TOTAL Trial for Severe Hypoplasia Investigators. Randomized Trial of Fetal Surgery for Severe Left Diaphragmatic Hernia. N Engl J Med. 2021 Jul 8;385(2):107-118. doi: 10.1056/NEJMoa2027030. Epub 2021 Jun 8. PMID 34106556
- See also: opens only end 2010 — http://www.totaltrial.eu